CLINICAL TRIAL: NCT02450916
Title: An Interview Study With Injured Workers Concerning Their Experiences With the Social
Brief Title: An Interview Study With Injured Workers Concerning Their Experiences With the Social Systems and Psychosocial Health Consequences
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201406016RINC
Record Dates: First submitted 2015-05-13; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Work-related Injury; Occupational Disease; Workers' Compensation; Psychological; Policy
Keywords: work-related injury; occupational disease; workers' compensation; psychological; policy
MeSH Terms: conditions — Occupational Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: In addition to physical discomforts, work-related injuries and illnesses often result in various forms of hardships, including economic hardship, labor conflicts and legal disputes. The physical and psychological health conditions are likely to be worsen when the social supporting systems are not well functioning. In this study, the investigators aim to conduct in-depth interviews with injured workers to study their experiences with the social systems, including employment protection system, workers' compensation system, health care system and other social welfare systems, and to explore how the systems may affect workers' physical and psychological health.

Methods: Face-to-face interviews will be conducted with a semi-structured questionnaire. Subjects who had ever experienced work-related injuries or diseases (including muscular skeletal disorders and work-related cardiovascular or cerebrovascular diseases) over the past 3 years are invited. The investigators anticipate to recruit a total of 60~100 cases, whom will be recruited through the assistance of occupational physicians, occupational health centers, labor groups and unions. Interview time will be limited to 1 hour.

Anticipated results and contribution: Findings of this study will help to advance our knowledge concerning the functions of current social systems and the hardships of workers who suffer from work-related injuries and diseases. Suggestions will be provided for the improvements of current systems.

Keywords: work-related injury, occupational disease, workers' compensation, psychological, policy.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who had ever experienced work-related injuries or diseases over the past 3 years are invited.
  Inclusion Criteria:
  1. work-related injuries
  2. work-related diseases
  Exclusion Criteria:
  1.transportation-related injuries on the way to work or on duty at work
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
self-rated mental health | 12 months after occupational injury or diseases
  using BSRS-5 scale
self-rated health | 12 months after occupational injury or diseases
  Self-rated health measured by a single question such as "in general, would you say that your health is excellent, very good, good, fair, or poor?" and a survey questionnaire in which participants assess different dimensions of their own health. This survey technique is commonly used in health research for its ease of use and its power in measuring health.

CONTACTS AND LOCATIONS:
Overall Officials: Yawen Cheng, Principal Investigator — Institute of Health Policy and Management, National Taiwan University, Taipei, Taiwan.
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan